CLINICAL TRIAL: NCT05772325
Title: The Effect of Brief Versus Individually Tailored Dietary Advice on Change in Lipids, Blood Pressure, and Diet in Patients With Inflammatory Joint Disease "The Diet Study"
Brief Title: The Effect of Brief Versus Individually Tailored Dietary Advice on Change in Lipids, Blood Pressure, and Diet in Patients With Inflammatory Joint Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University Hospital, Umeå (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol 03 02 23
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief standardized dietary advice (Active Comparator): The brief standardized 4-minute heart healthy dietary advice will be provided by an experienced cardiologist or rheumatologists.
  Interventions: Other: The brief standardized 4-minute heart healthy dietary advice
- Individually tailored diet counseling (Experimental): Participants in the intervention group will receive a 60 min individually tailored heart-friendly diet consultation by a dietitian.
  Interventions: Other: Individually tailored diet counseling

INTERVENTIONS:
Other: Individually tailored diet counseling — Participants in the intervention group will receive a 60 min individually tailored heart-friendly diet consultation by a dietitian
  Arms: Individually tailored diet counseling
Other: The brief standardized 4-minute heart healthy dietary advice — The brief standardized 4-minute heart healthy dietary advice will be provided by an experienced cardiologist or rheumatologists
  Arms: Brief standardized dietary advice

SUMMARY:
A randomized controlled study comparing brief dietary intervention with a personal, tailored dietary advice (60 min) on change in LDL-c and change in diet.

DETAILED DESCRIPTION:
Patients with inflammatory joint diseases (IJD) as rheumatoid arthritis (RA), spondylo arthropathy (SpA) and psoriatic arthritis (PsA) are at high risk of atherosclerotic cardiovascular disease. International recommendations for the prevention of cardiovascular disease recommend smoking cessation, physical activity, and dietary changes as part of treatment. Despite the evidence that behavioral counseling reduces overall cardiovascular risk, it is often an overlooked and underemphasized by clinicians. As of today, there is a knowledge gap regarding the efficacy of less intensive counseling sessions needed to obtain changes in dietary habits and clinical effects on CVD risk factors. Therefore, a brief dietary advice would be preferable if it could give a positive change in dietary habits and cholesterol. We have previously shown in a pilot study (8) that a 4 min. brief advice compared to a 60 min. personal tailored advice by a dietician on heart-friendly diet gave a similar change in dietary habits and LDL-c after 8 weeks in patients with IJD. The aim of the Diet Study is to perform a randomized controlled study comparing brief intervention (4 min) with a personal tailored dietary advice (60 min) on change in LDL-c and change in diet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either RA, PsA, or AS, between 30-80 years with an increased risk of future CVD, estimated using the CVD risk calculator. i.e. any risk > 5 -10 % predicted by Systematic Coronary Risk Evaluation (SCORE2) algorithm. Also, patients with very high risk (predicted risk >10%) as well as established atherosclerotic CVD (ASCVD) including previous myocardial infarction, coronary intervention (coronary artery bypass grafting or percutaneous coronary intervention), transient ischemic attack/strokes, atherosclerotic diseases of arteries as in the carotid artery or peripheral arterial disease (PAD) will also be included.

Exclusion Criteria:

1. Heart failure with systolic EF<40%
2. Kidney failure with GFR < 35
3. Liver failure
4. Mental disorder rendering the patient unable to comply with the protocol
5. Being able to speak the language of the country
6. Reduced cognitive function
7. Substance abuse

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
LDL cholesterol change from baseline | 8 weeks
  LDL cholesterol change from baseline

SECONDARY OUTCOMES:
Change in Healthy Diet Score (HDS) according to SmartDiet score | 8 weeks
  A self-administered 15-item food-frequency questionnaire (SmartDiet™) will be applied to assess subjects' average intake of: dairy products, mayonnaise products, meat, grain, fish, fruit, vegetables and snacks. The questionnaire has three response categories: Least healthy (1 point), Medium healthy (2 points) and Most healthy (3 points). The scores on the 15 questions are summed to obtain a Healthy Diet Score (HDS) ranging from 15 (worst) to 45 points (best). A change in the sum score of > 3 is considered a (clinical) significant change in diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No